CLINICAL TRIAL: NCT04023513
Title: Effects of Low or High Amounts of Dietary Protein and Resistance Training on Community-dwelling Older Adults: a Randomized Controlled Trial
Brief Title: Dietary Protein and Resistance Exercise in Elderly
Acronym: NUTRIAGINGPROT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Karl-Heinz Wagner, Professor of Human Nutrition, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FA219002
Record Dates: First submitted 2019-06-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Aging
Keywords: aging; protein intake; reistance training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strength Training and Protein high (Experimental): 6 weeks of high protein intake (additional 1g/kg bw/d) followed by a 8 weeks resistance training (Progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the protein intake remains.
  Interventions: Other: High protein intake; Other: Strength training
- Strength Training and Protein low (Experimental): 6 weeks of low protein intake (1g/kg bw/d) followed by a 8 weeks resistance training (Progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the protein intake remains.
  Interventions: Other: Low protein intake; Other: Strength training
- Control (Other): No Intervention.
  Interventions: Other: Control, no intervention

INTERVENTIONS:
Other: High protein intake — 6 weeks of high protein intake mainly via food (additional 1g/kg bw/d) followed by a 8 weeks resistance training (Progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the protein intake remains.
  Arms: Strength Training and Protein high
Other: Control, no intervention — No Intervention, control
  Arms: Control
Other: Low protein intake — 6 weeks of low protein intake (1g/kg bw/d) followed by a 8 weeks resistance training (Progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the protein intake remains
  Arms: Strength Training and Protein low
Other: Strength training — 6 weeks of different protein intake followed by a 8 weeks resistance training (Progressive strength training in a fitness center is applied; the intensity is adjusted continuously in order to obtain a sufficient training stimulus). During the training period the protein intake remains
  Arms: Strength Training and Protein high; Strength Training and Protein low

SUMMARY:
The aim of this randomized, observer-blind, controlled intervention study with parallel groups is to study the effect of resistance training (2x/week for 8 weeks) with and without different goals of protein intake on muscle strength, function and mass, oxidative stress parameters and the immune system in community dwelling persons.

Participants (n = 137) will be community-dwelling older adults. After a pre-participation screening participants will be distributed randomly but stratified by sex and age to one of the 3 groups (low protein + strength training, high protein + strength training, low protein and no strength training(=control)). Study participants are eligible if they are male or female with an age between 65 and 85 years and if their cognitive status as well as their physical fitness level allows to participate at the strength training sessions. Exclusion criteria comprise chronic diseases which contraindicate the training sessions, serious cardiovascular disease, diabetic retinopathy and manifest osteoporosis, a frailty index at or above 3, medication with anticoagulants or cortisone drugs and also regular strength training during the last six months.

Primary outcome measure is the change in the Chair Stand Test. Secondary outcome measures comprise anthropometric data, functional performance tests, immunological and oxidative stress parameters, microbiota, metabolomics, proteomics and the nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the age of 65 and 85 years of age
* Adequate mental condition in order to follow the instructions and to perform the resistance exercise independently (Mini-Mental-State >23)
* Independently mobile

Exclusion Criteria:

* Chronic diseases, which contraindicate a training participation
* Serious cardiovascular diseases (congestive chronic heart failure, severe or symptomatic aortic stenosis, unstable angina pectoris, untreated arterial hypertension, cardiac arrhythmias)
* Diabetic retinopathy
* Manifest osteoporosis
* Regular use of cortisone-containing drugs
* Regular strength training (> 1x / week) in the last 6 months before inclusion

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 137 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in chair stand test (repetitions) | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  The maximum number of completed cycles of unsupported chair rises (from a seated to a fully erected position (hip and knees straightened)) completed within 30 s is counted.

SECONDARY OUTCOMES:
Change from baseline in isometric quadriceps peak torque (Nm/kg) | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  Isokinetic peak torque measurements of knee extensors and flexors will be performed using a LIDO Multijoint II isokinetic loading dynamometer. Participants will be tested in a sitting posion with their hip flexed at approximately 90° and subjects securely strapped to the seat of the chair using adjustable trunk and waist stabilisation belts. The anatomic axis of the knee rotation at the knee joint will aligned with the machine axis of rotation to insure similar movements for all participants. Two continuous maximal repetitions of knee extensors and knee flexors will be performed concentrically at each angular velocity (60°/s and 120°/s) for peak torque recording.
Change from baseline in handgrip strength (kg) | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  Handgrip strength of the right hand will be measured to the nearest kilogram (kg) using a hand Dynamometer. Participants will be encouraged to perform a maximal contraction within approximately 4 to 5 s. After a rest of 60 s, participants will be asked to perform a second trial. The highest score of maximum voluntary contraction will be used for data analyses.
Change from baseline in muscle mass with BIA (kg) | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
Change from baseline in 6min walking test (distance in meter) | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
Change from baseline in the composition of gut-microbiota | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  Gene sequencing of the 16S rRNA on the stool samples are performed to identify the microbes down to genus level, as well as the microbrobiota diversity and relative abundance.
Change from baseline in stool short-chain fatty acids (SCFAs) | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  The stool short-chain fatty acids (SCFAs) will be extracted and quantitatively analysed by gas chromatography.
Change from baseline in oxidative stress marker such as malondialdehyd | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  The investigators will consider changes in plasma concentrations of oxidative stress marker such as malondialdehyde from baseline to the end of the intervention.
Change from baseline in inflammatory marker (i.g. IL-6, TNF-alpha) | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  The investigators will consider changes in plasma concentrations of Interleukin 1 (IL-1), IL-6, IL-8, IL-10, TNF-alpha
Change from baseline in the metabolomics response | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  The metabolomic response (ie all metabolites) to the interventions will be analyzed using both nuclear magnetic resonance (NMR) and mass spectrometry (MS) techniques. Patterns of metabolites will be evaluated with statistical techniques, ie discriminant analysis and principal component analysis.
Change from baseline in the amino acid pattern | baseline, after dietary intervention (6 weeks) and after dietary and strength training (14 weeks)
  The plasma amino acid pattern will be assessed with HPLC-MS.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Department of Nutritional Sciences, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spahits H, Unterberger S, Aschauer R, Zohrer PA, Draxler A, Franzke B, Strasser EM, Wessner B, Wagner KH, Tahir A. Impact of a high-protein diet with and without strength training over 17 weeks on the plasma metabolome in older adults. Age Ageing. 2026 Feb 1;55(2):afag010. doi: 10.1093/ageing/afag010. PMID 41638233
- [Derived] Franzke B, Bileck A, Unterberger S, Aschauer R, Zohrer PA, Draxler A, Strasser EM, Wessner B, Gerner C, Wagner KH. The plasma proteome is favorably modified by a high protein diet but not by additional resistance training in older adults: A 17-week randomized controlled trial. Front Nutr. 2022 Aug 5;9:925450. doi: 10.3389/fnut.2022.925450. eCollection 2022. PMID 35990326
- [Derived] Unterberger S, Aschauer R, Zohrer PA, Draxler A, Franzke B, Strasser EM, Wagner KH, Wessner B. Effects of an increased habitual dietary protein intake followed by resistance training on fitness, muscle quality and body composition of seniors: A randomised controlled trial. Clin Nutr. 2022 May;41(5):1034-1045. doi: 10.1016/j.clnu.2022.02.017. Epub 2022 Feb 24. PMID 35390727